CLINICAL TRIAL: NCT01047969
Title: Non-Operative Treatment for Rectal Cancer Following Complete Response to Neo-Adjuvant Therapy
Brief Title: Avoiding Surgery in Rectal Cancer After Pre-Operative Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ann Gandolfi, Julie Curtis, Royal Marsden NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2759
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2016-05

CONDITIONS: Rectal Adenocarcinoma
Keywords: locally invasive high-risk rectal adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemotherapy, Adjuvant; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Adjuvant Chemotherapy — If after MRI + FDG-PET 8 weeks post CRT the patient shows no visible tumour or further regression adjuvant chemotherapy will be considered.
Procedure: Surgery — If after MRI + FDG-PET 8 weeks post CRF no further regression or growth of disease occurs the patient will be referred for surgery.

SUMMARY:
The objective of Timing and Deferral of Rectal Surgery Following a Continued Response to Pre-operative CRT study is to establish the time to maximum tumour response following CRT, and to investigate whether surgery can be safely avoided within the tight framework of the trial follow-up protocol in a small group of patients where the cancer becomes undetectable by imaging modalities.

DETAILED DESCRIPTION:
The study uses MRI in combination with FDG-PET CT and clinical examination (tri-modality assessment) to assess for a continued incremental response to CRT. Surgery is NOT withheld from patients entering this study. Indeed, surgery is an option at each stage of patient follow-up and is a crucial component of a patient's treatment pathway should no further regression of disease be detected through stringent follow-up. If a status of 'no detectable disease' by serial MRI, CT-PET and clinical assessment is achieved and the patient wishes not to have surgery, they will continue to be carefully monitored within the framework of the trial follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Locally invasive high-risk rectal adenocarcinoma as defined by the presence on MRI of at least one of the following: i) Tumours within 1mm of mesorectal fascia i.e. circumferential resection margin threatened or involved ii)T3 tumours at/below levators iii)Tumours extending ≥5mm into peri-rectal fat iv)T4 tumours (including the involvement of bladder or vagina if surgical resection is possible with clear margins) v)Presence of extra-mural venous invasion (primary tumour is therefore at least T3) vi)T2 N0/1/2 tumours requiring Abdomino-Perineal Excision, within 1mm of mesorectal fascia i.e. circumferential resection margin threatened or involved
* The absence of malignant pelvic side-wall disease, local recurrence (either after TME or wide local excision) or metastatic disease
* Completion of pre-operative long-course CRT
* No viable disease seen at MRI performed 4 weeks after long-course CRT, confirmed at 8 week MRI
* Evidence of partial response of rectal tumour to pre-operative long-course CRT at 4 week MRI which continues to show an incremental response at 8 week MRI.
* Histological diagnosis of adenocarcinoma of rectum.
* WHO performance status 0, 1 or 2.
* No evidence of metastatic disease as determined by CT scan of chest, abdomen, pelvis or other investigations such as PET scan or biopsy if required.
* Informed written consent

Exclusion Criteria:

* Age < 18 years.
* Absence of concomitant chemotherapy.
* RT dose below 50Gy.
* Stable disease at 4 week MRI.
* Disease that demonstrates a partial response at 4 week MRI but shows no evidence of an incremental response at 8 week MRI.
* Pregnancy or breast feeding
* Short course pre-operative radiotherapy
* Previous pelvic radiotherapy
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Any contra-indication to MRI scanning, eg Cardiac Pacemaker or Hip prosthesis.
* Any patients within the EXPERT-C trial.
* Tumours which are mucinous (>50% mucin seen on MRI), as these are more likely to be PET negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-06-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
To estimate the percentage of patients who can safely omit surgery, defined as the percentage of patients at two years after end of CRT who have not had surgery and who are in CR (no detectable local disease) | Two years post end of chemoradiotherapy
To prove the safety of deferred surgery, as measured by the percentage of patients who have local failure at two years, where local failure is defined as positive margin status of resected tumour or surgically unsalvageable disease. | Two years post end of chemoradiotherapy

SECONDARY OUTCOMES:
Time to distant disease | The time to the first diagnosis of lymph node or other distant disease, confirmed via PET/CT, MRI, CT or pathology
Time to maximal tumour response after CRT | The time when tumour regressed to its minimum thickness and when MRI
Time to local re-growth | The time until the first recorded increase in Mandard grade, or tumour thickness or length, on MRI
Percentages of positive margins, and sphincter-preservation rates in patients who have had surgery | At the end of the study - all patients who had surgery for progression of local disease
Progression-free and overall survival | Measured from the end of CRT (cohort A) or end of adjuvant chemotherapy (cohort B). Surviving patients in continued CR will be censored at the date of last follow-up (clinic visit or imaging).
Quality of Life including long-term bowel, urinary and sexual function | 10 years after registration, or five years post-surgery.
To correlate the expression of biological markers which may predict for pathological complete response with progression free survival | End of study

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden NHS Foundation Trust, London, United Kingdom